CLINICAL TRIAL: NCT04804423
Title: Evaluation of the Efficacy of Fluoride Therapies on Hypersensitive Carious Lesions in Primary Teeth
Brief Title: Fluoride Therapies on Hypersensitive Carious Lesions in Primary Teeth
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: SDI Limited (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID-KinderZZMK-2020
Record Dates: First submitted 2021-03-04; First posted 2021-03-18 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Dentin Hypersensitivity; Active Dental Caries
MeSH Terms: conditions — Dentin Sensitivity | interventions — silver fluoride; sodium fluoride topical preparation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluoride varnish (Duraphat®) (Active Comparator): Fluoride varnish application is recommended by the German National Health System for managing hypersensitivity and dental caries. Sodium fluoride varnish (Duraphat®) will be applied on hypersensitive active carious lesions (ICDAS 5).
  Interventions: Drug: Sodium fluoride varnish (generic name; Duraphat®)
- Silver fluoride and potassium iodide (Riva Star®) (Experimental): Silver fluoride and potassium iodide (Riva Star®) is primarily indicated for relieving hypersensitivity will be applied on hypersensitive active carious lesions (ICDAS 5) following isolation of the affected teeth and according to manufacturer's instructions.
  Interventions: Drug: 38% Silver Fluoride and Potassium Iodide solution (generic name; Riva Star®)

INTERVENTIONS:
Drug: 38% Silver Fluoride and Potassium Iodide solution (generic name; Riva Star®) — 38% silver fluoride will be applied to the surface of the isolated hypersensitive carious lesion followed by application of potassium iodide solution and according to manufacturer's instructions.
  Other Names: Riva Star®
  Arms: Silver fluoride and potassium iodide (Riva Star®)
Drug: Sodium fluoride varnish (generic name; Duraphat®) — 22,600 ppm sodium fluoride varnish will be applied on the surface of the affected hypersensitive active carious lesions.
  Other Names: Duraphat®
  Arms: Fluoride varnish (Duraphat®)

SUMMARY:
This observational cohort study aims to evaluate the short-term (3 months) efficacy of the standard fluoride therapy in the German National Health System for managing hypersensitive carious lesions in primary teeth (fluoride varnish application), and further compare it to a different fluoride therapy utilizing a silver-containing fluoride agent combined with potassium iodide solution.

DETAILED DESCRIPTION:
A single trained investigator will screen for possible study participants of children aged 2-5 years old, and their parents will be asked to participate in the study. The participants will be consecutively recruited from regular clinic attendees of the Department of Preventive and Pediatric Dentistry at the University of Greifswald, from whom present with active carious lesions (ICDAS 5) along symptoms of hypersensitivity to be treated with fluoride varnish, and further compared to participants treated with silver fluoride and potassium iodide application.

Eligibility to the study will be determined by a single trained examiner through clinical findings of caries activity according to Bjørndal criteria, and reported history of hypersensitivity symptoms obtained from the parent/caregiver of the participant, followed by hypersensitivity confirmatory test using a triple syringe air blast on the exposed surface of the carious lesion to allocate areas with suspected dentin hypersensitivity.

After clinical examination and obtainment of an informed consent, eligible children will be treated with fluoride varnish application (Duraphat®), or silver fluoride and potassium iodide application (Riva Star®) according to manufacturer's instructions.The participant's behavior shall be evaluated at the beginning, during and after treatment. Plaque Index (API) and Papillary Bleeding Index (PBI) will also be assessed prior to treatment and at the 3-months mark. Procedures will be performed by six different dentists (four pediatric specialists and two post-graduate pediatric dentistry students), all of whom were briefed on the study protocol and received instructions in carrying in the interventions according to the manufacturer's guide, and their technical opinions regarding the performed procedures will be obtained following the procedure. Follow up examinations after 3 months will be done by a single examiner. Only one tooth per child will be included in the analysis.

Data and information of this study will be recorded, handled, and stored in an organized and secure way, to allow its accurate reporting, interpretation, and verification. To assure confidentiality of clinical records, an unambiguous subject identification code will be used. Patients who are no longer willing to continue in the study will have the right to quit at any time without any penalty.

All variables will be statistically analyzed using descriptive statistics, plots, and tests of normality. Means and standard deviations (SD) will be calculated for all quantitative variables, while frequencies and percentages will be calculated for categorical variables.

Comparison between the two study groups will utilize independent samples t-test for quantitative normally distributed variables, and Mann-Whitney U for quantitative non-normally distributed variables and qualitative ordinal variables. Chi-squared and Fisher exact tests will be performed for comparing qualitative nominal variables between the two study groups. Comparing the baseline and follow-up shall be done using paired t-test when the variable is normally distributed, and Wilcoxon signed rank test when the variable is not normally distributed. For comparing lesion activity before and after treatment, McNemar test will be used and Friedman test for comparing the children's behavior at 3 different time points (before, during and after treatment).

A Significance will be set at p<0.05. Data will be analyzed using IBM SPSS statistical software for windows (version 25).

ELIGIBILITY:
Inclusion Criteria:

* Reported hypersensitivity in primary teeth associated with the presence of active carious lesions (ICDAS 5).
* Healthy children aged 2-5 years.
* Not using any desensitizer for 1-month prior the study.
* Willing to be examined.

Exclusion Criteria:

* Previously restored teeth.
* Teeth with signs or symptoms of irreversible pulpitis.
* Patients with any systemic disease requiring special considerations during their dental treatment.
* Parents/children who declined to participate in the study.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Hypersensitivity pain relief | 3 Months
  The degree of pain severity will be quantified by a visual analogue scale - VAS; 0-10, ranging across a continuum from none (0) to a severe amount of pain (10).

SECONDARY OUTCOMES:
Activity of carious lesions | 3 Months
  Lesions will be assessed for caries activity using visual tactile criteria (Bjørndal Criteria; 0 - 9= sound -missing tooth) 0. Sound
  1. Active lesion in enamel , without cavity ( bright surface with brown discoloration )
  2. Active cavity in enamel ( opaque enamel surface and loss of substance )
  3. Active cavity in enamel ( bright surface , brown discoloration, wet dentin )
  4. Inactive cavity in enamel ( bright surface, brown discoloration and loss of substance )
  5. Active cavity in enamel/dentin ( yellow or light brown discoloration , wet dentin )
  6. Inactive cavity in enamel/dentin ( dark brown discoloration, hard and dry dentin )
  7. Pulpal involvement or root stumps
  8. Filled tooth
  9. Missing tooth
Patient Acceptance | Only at baseline (begining, during and after procedure)
  Children's behavior before, during and after treatment was assessed using Frankl's Scale
  1. Definitely positive: Good rapport with the dentist, interested in the dental procedure, laughing and enjoying the situation
  2. Positive: Acceptance of treatment; at time cautious, willingness to comply with the dentist, at times with reservation but patient follows the dentist's directions cooperatively
  3. Negative: Reluctant to accept treatment; uncooperative, some evidence of negative attitude but not pronounced
  4. Definitely negative: Refusal of treatment, crying forcefully, fearful, or any other overt evidence of extreme negativism
Operating Dentists' Opinion About the Procedure Performed | Will be recorded immediately after the procedure
  Dentist's technical opinion regarding the procedures and materials used in the study groups will be collected directly after performing the procedure using 5-point Likert scales.

OTHER OUTCOMES:
O'Leary Plaque Control Index | 3 Months
  Visual assessment of plaque covered surfaces following application of a disclosing solution. The number of positively scored surfaces is divided by the total number of tooth surfaces evaluated, and the result is multiplied by 100 to express the index as a percentage
  O'Leary Palque Index will be clinically evaluated prior to treatment and at the 3-months follow up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed H Abudrya, BDS, MSc., Principal Investigator — The Department of Preventive and Pediatric Dentistry, University of Greifswald
Locations (1):
- The Department of Preventive and Pediatric Dentistry, University of Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] West N, Seong J, Davies M. Dentine hypersensitivity. Monogr Oral Sci. 2014;25:108-22. doi: 10.1159/000360749. Epub 2014 Jun 26. PMID 24993261
- [Background] Crystal YO, Janal MN, Hamilton DS, Niederman R. Parental perceptions and acceptance of silver diamine fluoride staining. J Am Dent Assoc. 2017 Jul;148(7):510-518.e4. doi: 10.1016/j.adaj.2017.03.013. Epub 2017 Apr 27. PMID 28457477
- [Background] Use of Silver Diamine Fluoride for Dental Caries Management in Children and Adolescents, Including Those with Special Health Care Needs. Pediatr Dent. 2018 Oct 15;40(6):152-161. PMID 32074885
- [Background] Gao SS, Zhang S, Mei ML, Lo EC, Chu CH. Caries remineralisation and arresting effect in children by professionally applied fluoride treatment - a systematic review. BMC Oral Health. 2016 Feb 1;16:12. doi: 10.1186/s12903-016-0171-6. PMID 26831727
- [Background] Machiulskiene V, Campus G, Carvalho JC, Dige I, Ekstrand KR, Jablonski-Momeni A, Maltz M, Manton DJ, Martignon S, Martinez-Mier EA, Pitts NB, Schulte AG, Splieth CH, Tenuta LMA, Ferreira Zandona A, Nyvad B. Terminology of Dental Caries and Dental Caries Management: Consensus Report of a Workshop Organized by ORCA and Cariology Research Group of IADR. Caries Res. 2020;54(1):7-14. doi: 10.1159/000503309. Epub 2019 Oct 7. PMID 31590168
- [Background] Poulsen S, Errboe M, Hovgaard O, Worthington HW. Potassium nitrate toothpaste for dentine hypersensitivity. Cochrane Database Syst Rev. 2001;(2):CD001476. doi: 10.1002/14651858.CD001476. PMID 11405992
- [Background] Splieth CH, Tachou A. Epidemiology of dentin hypersensitivity. Clin Oral Investig. 2013 Mar;17 Suppl 1(Suppl 1):S3-8. doi: 10.1007/s00784-012-0889-8. Epub 2012 Dec 7. PMID 23224064
- [Background] Santamaria RM, Innes NPT, Machiulskiene V, Schmoeckel J, Alkilzy M, Splieth CH. Alternative Caries Management Options for Primary Molars: 2.5-Year Outcomes of a Randomised Clinical Trial. Caries Res. 2017;51(6):605-614. doi: 10.1159/000477855. Epub 2017 Dec 20. PMID 29258064
- [Background] Santamaria RM, Abudrya MH, Gul G, Mourad MS, Gomez GF, Zandona AGF. How to Intervene in the Caries Process: Dentin Caries in Primary Teeth. Caries Res. 2020;54(4):306-323. doi: 10.1159/000508899. Epub 2020 Aug 27. PMID 32854105
- See also: DA: Food and Drug Administration. Diammine Silver Fluoride Dental Hypersensitivity Varnish. — http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm?ID=K102973